CLINICAL TRIAL: NCT03060941
Title: Promoting Activity in Cancer Survivors
Acronym: PACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 092016-004
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Physical Activity; Breast Cancer
MeSH Terms: conditions — Motor Activity; Breast Neoplasms | interventions — Architectural Accessibility

STUDY DESIGN:
Intervention Model Description: The 500 participants in the physical activity intervention will be randomly assigned to one of sixteen intervention groups (see Table below). Randomization will be stratified by clinical site. The randomization scheme will be conducted by the study statistician. The randomization scheme will consist of balanced blocks within each stratum, with block size will be varied and randomly permuted. Allocation will occur following completion of baseline assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Group 1 (Experimental): Physical activity education
  Interventions: Behavioral: Physical activity education
- Group 2 (Experimental): Physical activity education and facility access
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access
- Group 3 (Experimental): Physical activity education and supervised exercise sessions
  Interventions: Behavioral: Physical activity education; Behavioral: Supervised exercise sessions
- Group 4 (Experimental): Physical activity education and self-monitoring (Fitbit)
  Interventions: Behavioral: Physical activity education; Behavioral: Self-monitoring (Fitbit)
- Group 5 (Experimental): Physical activity education and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Active living counseling
- Group 6 (Experimental): Physical activity education, facility access, and supervised exercise sessions
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Supervised exercise sessions
- Group 7 (Experimental): Physical activity education, facility access, and self-monitoring (Fitbit)
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Self-monitoring (Fitbit)
- Group 8 (Experimental): Physical activity education, facility access, and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Active living counseling
- Group 9 (Experimental): Physical activity education, supervised exercise sessions, and self-monitoring (Fitbit)
  Interventions: Behavioral: Physical activity education; Behavioral: Supervised exercise sessions; Behavioral: Self-monitoring (Fitbit)
- Group 10 (Experimental): Physical activity education, supervised exercise sessions, and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Supervised exercise sessions; Behavioral: Active living counseling
- Group 11 (Experimental): Physical activity education, self-monitoring (Fitbit), and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Self-monitoring (Fitbit); Behavioral: Active living counseling
- Group 12 (Experimental): Physical activity education, facility access, supervised exercise sessions, and self-monitoring (Fitbit)
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Supervised exercise sessions; Behavioral: Self-monitoring (Fitbit)
- Group 13 (Experimental): Physical activity education, facility access, supervised exercise sessions, and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Supervised exercise sessions; Behavioral: Active living counseling
- Group 14 (Experimental): Physical activity education, facility access, self-monitoring (Fitbit), and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Self-monitoring (Fitbit); Behavioral: Active living counseling
- Group 15 (Experimental): Physical activity education, supervised exercise sessions, self-monitoring (Fitbit), and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Supervised exercise sessions; Behavioral: Self-monitoring (Fitbit); Behavioral: Active living counseling
- Group 16 (Experimental): Physical activity education, facility access, supervised exercise sessions, self-monitoring (Fitbit), and active living counseling
  Interventions: Behavioral: Physical activity education; Behavioral: Facility access; Behavioral: Supervised exercise sessions; Behavioral: Self-monitoring (Fitbit); Behavioral: Active living counseling

INTERVENTIONS:
Behavioral: Physical activity education — Participants will be given educational materials on how to increase physical activity levels.
Behavioral: Facility access — Participants will receive at 6 month membership to a local fitness facility.
  Arms: Group 12; Group 13; Group 14; Group 16; Group 2; Group 6; Group 7; Group 8
Behavioral: Supervised exercise sessions — Participants will attend weekly supervised exercise sessions with an exercise interventionist.
  Arms: Group 10; Group 12; Group 13; Group 15; Group 16; Group 3; Group 6; Group 9
Behavioral: Self-monitoring (Fitbit) — Participants will be given a Fitbit to monitor their physical activity levels.
  Arms: Group 11; Group 12; Group 14; Group 15; Group 16; Group 4; Group 7; Group 9
Behavioral: Active living counseling — Participants will attend 12 biweekly educational sessions about how to increase their physical activity levels.
  Arms: Group 10; Group 11; Group 13; Group 14; Group 15; Group 16; Group 5; Group 8

SUMMARY:
A randomized multi-component physical activity intervention for breast cancer survivors.

DETAILED DESCRIPTION:
The research project is a study to assess the effects of a multi-component intervention in increasing physical activity among breast cancer survivors. Individuals meeting inclusion/exclusion criteria will be randomized to one of sixteen intervention groups for the 6 months. Intervention components will include print-based education, self-monitoring, Active Living counseling, supervised exercise sessions, and facility access. Blood samples will be collected at baseline. Assessments (anxiety, stress, sleep) and sample collection will also occur at 3 time points during the intervention (Weeks 13 and 25). Changes in physical activity will be assessed for each intervention group.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer survivors between 3 months and 5 years post-treatment
* report <150 minutes of moderate-to-vigorous physical activity (MVPA) on the GPAQ
* physically able to engage in physical activity

Exclusion Criteria:

* medical condition contraindicating physical activity participation
* cognitively unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity measured by Actigraph accelerometer | 24 weeks
  Measure physical activity at baseline and follow-up periods (3- and 6-months post-baseline) and assess percentage of survivors meeting physical activity guideline recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, MD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rethorst CD, Carmody TJ, Argenbright KE, Mayes TL, Hamann HA, Trivedi MH. Considering depression as a secondary outcome in the optimization of physical activity interventions for breast cancer survivors in the PACES trial: a factorial randomized controlled trial. Int J Behav Nutr Phys Act. 2023 Apr 20;20(1):47. doi: 10.1186/s12966-023-01437-x. PMID 37081460
- [Derived] Rethorst CD, Hamann HA, Carmody TJ, Sharp KJ, Argenbright KE, Haley BB, Skinner CS, Trivedi MH. The Promoting Activity in Cancer Survivors (PACES) trial: a multiphase optimization of strategy approach to increasing physical activity in breast cancer survivors. BMC Cancer. 2018 Jul 18;18(1):744. doi: 10.1186/s12885-018-4662-5. PMID 30021554